CLINICAL TRIAL: NCT02630901
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study of PRX003 Administered by Intravenous Infusion in Subjects With Psoriasis
Brief Title: Multiple Ascending Dose Study of PRX003 in Subjects With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRX003-102
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2016-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRX003 (Experimental)
  Interventions: Drug: PRX003
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PRX003
  Arms: PRX003
Other: Placebo
  Arms: Placebo

SUMMARY:
This multiple ascending dose study is to determine safety, tolerability, pharmacokinetics and immunogenicity of PRX003 in approximately 56 patients with Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 80 years of age (inclusive), body weight range of ≥ 45 kg (99 lbs) to ≤ 120 kg (264 lbs) and a body mass index (BMI) of 18 - 35 kg/m2
2. Provide written informed consent
3. PASI score of ≥12
4. Plaque psoriasis covering ≥10% of BSA
5. s-PGA score of 3 or 4
6. Able to perform all protocol-specified assessments and comply with the study visit schedule
7. Female subjects who are not postmenopausal or surgically sterile must use physician approved contraception for at least 60 days prior to Baseline (Day 1/Visit 2) to 12 weeks following the last study drug administration. Unless they are at least 2 years postmenopausal or surgically sterile, women must have a pregnancy test with follicle stimulating hormone (FSH) >40 IU/L and estradiol <20 pg/mL (unless on hormone-replacement therapy). Women of childbearing potential must be non lactating and have a negative serum pregnancy test (beta human chorionic gonadotropin [β HCG]) at Screening (Visit 1).
8. If male, must be surgically sterile or must agree to use physician-approved contraception from Baseline (Day 1/Visit 2) to 12 weeks following the last study drug administration

Exclusion Criteria:

1. Presents with psoriasis that is predominantly guttate, erythrodermic, inverse, pustular or palmo-plantar, or an unstable form of psoriasis
2. Receipt of any of the following within the specified time frame prior to Baseline (Day 1/Visit 2):

   * Topical psoriasis treatments (other than low-potency topical corticosteroids or emollients, which are permitted during the study) within 2 weeks
   * Systemic (nonbiologic) psoriasis treatments within 4 weeks or 5 half-lives (whichever is longer)
   * Biologic psoriasis treatments within 12 weeks or 5 half-lives (whichever is longer)
   * Drugs that appear to have a strong causal relationship to psoriasis (e.g., beta-blockers and lithium) within 4 weeks or 5 half-lives (whichever is longer)
   * Phototherapy within 4 weeks
3. Participation in recreational sunbathing or use of a sun-bed (e.g., tanning salon) within 7 days prior to Baseline (Day 1)
4. Any major medical illness or unstable medical condition that, in the opinion of the Investigator or Sponsor, may interfere with the subject's ability to comply with study procedures or abide by study restrictions, or with the ability to interpret safety data, including, but not limited to:

   * Within 5 years of Screening (Visit 1)
   * History of cancer with the exception of fully excised non-melanoma skin cancer
   * History of stroke
   * History of epilepsy or seizure disorder other than febrile seizures as a child, or any seizure or loss of consciousness
   * History of or active autoimmune disease (other than psoriasis or PsA)
   * Within 2 years of Screening (Visit 1)
   * Myocardial infarction
   * Clinically significant cardiovascular disease including any of the following: unstable angina, decompensated congestive heart failure, clinically significant arrhythmias
   * Vascular diseases, including, but not limited to, blood clotting disorders, atherosclerosis, aneurysms, and renal artery disease
5. Hypotension (systolic blood pressure [BP] ≤85 millimeters of mercury [mmHg]) at Baseline (Day 1/Visit 2) predose or a known history or documentation of hypotension on more than one occasion within 3 months prior to Baseline (Day 1/Visit 2)
6. Uncontrolled hypertension as indicated by a resting systolic BP ≥150 mmHg or diastolic BP ≥95 mmHg at Screening (Visit 1) or Baseline (Day 1/Visit 2) predose or a known history or documentation of uncontrolled hypertension on more than one occasion within 3 months prior to Baseline (Day 1/Visit 2)
7. Clinically significant systemic infection (e.g., chronic or acute infection, urinary tract infection, upper respiratory infection) within 30 days of Baseline (Day 1/ Visit 2), or a history or presence of recurrent or chronic infection (e.g., viral infections [including hepatitis B or C, human immunodeficiency virus (HIV)], bacterial infections, systemic fungal infections, or syphilis)
8. History of any inflammatory bowel disease
9. Any current psychiatric diagnosis according to Diagnostic and Statistical Manual of Mental Disorders IV Text Revision (DSM-IV-TR) that may interfere with the subject's ability to perform the study and all assessments (e.g., alcohol or drug-related abuse or alcohol dependence, or alcohol or drug-related dementia, major depression, developmental disability, schizophrenia, bipolar disorder). Note: Subjects with adequately controlled depression for at least 6 months are not excluded; however, suicidal ideation or attempt at any time within the past year is exclusionary.
10. A positive tuberculosis skin test (TST) or a positive interferon-gamma release assay (IGRA) during Screening (Visit 1).

    Note: In the event a subject has had a TST or IGRA within 3 months before Baseline (Day 1/Visit 2), this does not need to be repeated during screening and the previous result can be carried forward and used in this study.

    Prior standard treatment for latent tuberculosis and prior exposure to tuberculosis with subsequent standard prophylactic treatment is allowed if recent (within ˂ 30 days) negative chest X-ray.
11. Any of the following laboratory abnormalities at Screening (Visit 1):

    * Total bilirubin (unless attributed to Gilbert's syndrome) >1.5 times the upper limit of normal (× ULN), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × ULN
    * Serum creatinine >133 µmol/L (1.5 mg/dL)
    * Hemoglobin <11.5 g/dL for males or <10.0 g/dL for females, absolute neutrophil count of ˂1500/µL (with the exception of a documented history of a chronic benign neutropenia), or platelet count of <120,000/µL
12. Use of an investigational product or device or participation in a drug research study within a period of 30 days (or 5 half-lives of the drug, whichever is longer) prior to Screening (Visit 1); for investigational products or drug research studies relating to psoriasis or arthritis, the duration will be extended to 12 weeks (or 5 half-lives of the drug, whichever is longer) prior to Screening (Visit 1)
13. Allergy to any of the components of PRX003 such as histidine, sucrose and polysorbate 20
14. Receipt of any vaccine (with the exception of seasonal influenza) within 30 days prior to Screening (Visit 1)
15. Donation of >500 mL of blood within 3 months prior to Screening (Visit 1)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as determined by number of subjects with adverse events | 6 months
Determination of pharmacokinetics parameters | 20 weeks
  time of the maximum measured concentration (Tmax)
Determination of pharmacokinetics parameters | 20 weeks
  area under the concentration-time curve from time zero to the last quantifiable concentration time-point (AUClast)
Determination of pharmacokinetics parameters | 20 weeks
  maximum concentration (Cmax)
Determination of pharmacokinetics parameters | 20 weeks
  area under the concentration-time curve from time zero extrapolated to infinity (AUCinf)
Determination of pharmacokinetics parameters | 20 weeks
  elimination rate constant
Determination of pharmacokinetics parameters | 20 weeks
  terminal elimination half life (t½)
Determination of pharmacokinetics parameters | 20 weeks
  clearance (CL)
Determination of pharmacokinetics parameters | 20 weeks
  apparent volume of distribution (Vd)
Determination of pharmacokinetics parameters | 20 weeks
  average concentration over a dosing interval (Cav)
Determination of pharmacokinetics parameters | 20 weeks
  area under the plasma concentration-time curve for a dosing interval (AUCtau)
Determination of pharmacokinetics parameters | 20 weeks
  minimum observed concentration (Cmin)

SECONDARY OUTCOMES:
Immunogenicity as determined by measurement of anti-PRX003 antibodies | 20 weeks
  antibody titers will be listed and summarized

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - TCR Medical Corporation, San Diego, California
  - Universal Medical and Research Center, LLC, Coral Gables, Florida
  - Renstar Medical Research, Ocala, Florida
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Virginia Clinical Research Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No